CLINICAL TRIAL: NCT02392143
Title: Promoting CRC Screening in a Hard-To-Reach, Low-Income Minority Population
Brief Title: Promoting CRC Screening in an Urban Minority Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Columbia University (Other); 1199SEIU Benefit and Pension Funds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 542376
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Printed Education Material (Active Comparator): Participants received printed education materials (PEM) sent by first class mail.
  Interventions: Other: Printed Education Material
- Academic Detailing (Active Comparator): Participants' primary care physicians (PCPs) received academic detailing (AD) to improve colorectal cancer screening referral and follow-up practices.
  Interventions: Other: Academic Detailing
- Academic Detailing+Telephone Education (Active Comparator): Participants' primary care physicians (PCPs) received academic detailing (AD) to improve colorectal cancer screening referral and follow-up practices and participants received tailored telephone education (TTE).
  Interventions: Other: Academic Detailing+Telephone Education

INTERVENTIONS:
Other: Printed Education Material — The printed education material described the importance of early detection and prevention, risk factors, and the importance of talking to your doctor about CRC screening. The PEM highlighted colonoscopy as being the only test that can identify and prevent CRC and described how to prepare for a colonoscopy beginning seven days prior to the test [18]. The PEM also described other CRC screening tests, including the FOBT, FIT, sigmoidoscopy, barium enema and virtual colonoscopy.
  Other Names: Print education
  Arms: Printed Education Material
Other: Academic Detailing — Academic detailing (AD) involved an in-person visit from a member of the research team who attempted to communicate strategies for improving CRC screening uptake in the practice's patient panel. A brief description of the RCT was followed by a semi-structured interview assessing usual practice regarding CRC screening referral and follow up. The direction of the discussion was guided by PCP responses. A variety of resources were provided. Specific directives were following up to make sure patients had made appointments with a gastroenterologist and offering home stool tests. The detailer attempted to elicit a verbal commitment to do at least one new thing to strengthen the probability that patients would be screened.
  Arms: Academic Detailing
Other: Academic Detailing+Telephone Education — PCPs received AD as described in the Academic Detailing arm. In addition, participants received tailored telephone education (TTE) which focused on identifying and addressing barriers that might impede screening. Verbal commitments were elicited to speak with their PCP and make an appointment for a colonoscopy, or request a home stool test, as appropriate. Follow-up calls assessed progress towards achieving goals.
  Other Names: Academic Detailing+Tailored Telephone Education
  Arms: Academic Detailing+Telephone Education

SUMMARY:
The purpose of this study (Healthy Colon Project II) is to evaluate different educational approaches for increasing rates of colorectal cancer (CRC) screening in a hard-to-reach urban minority population with health insurance.

DETAILED DESCRIPTION:
This project is an extension of the investigators' earlier study (Healthy Colon Project I) in which the investigators demonstrated that telephone outreach to individuals had a significant effect on CRC screening in a hard-to-reach, working class, urban minority population (~27.0% screened who received telephone outreach vs. ~6.1% screened who received printed educational materials). Additional investigation suggested the possible benefits of intervening with primary care physicians (PCPs) regarding their CRC screening referral and follow-up practices.

In the current project, the investigators conducted a 3-group randomized trial. The aims are as follows: Aim 1: Evaluate the incremental effect of tailored telephone education (TTE), over and above the effect of academic detailing (AD), for increasing rates of CRC screening 12-months post-randomization; Aim 2: Evaluate the effect of academic detailing alone (AD) over minimal intervention (control group), for increasing rates of CRC screening 12-months post-randomization; Aim 3: Identify factors that mediate the effectiveness of the interventions; and Aim 4: Identify factors that moderate the effectiveness of the interventions among subgroups.

In one group, participants received printed education materials. In a second group, participants' PCPs received academic detailing (AD) to improve CRC screening referral and follow-up practices. And in a third group, PCPs received AD and participants received tailored telephone education (TTE). Participants were members of a union-based, self-administered and self-insured benefit fund in the NYC metropolitan area.

The educational intervention approaches were informed by the investigators' earlier study among this population, with the goal of helping participants to make an informed choice about screening. The CRC PEM described the importance of early detection and prevention, risk factors, and the importance of talking to the subject's doctor about CRC screening. The PEM highlighted colonoscopy as being the only test that can identify and prevent CRC and described how to prepare for a colonoscopy beginning seven days prior to the test. The PEM also described other CRC screening tests, including the FOBT, FIT, sigmoidoscopy, barium enema and virtual colonoscopy. Academic detailing (AD) involved an in-person visit from a member of the research team who attempted to communicate strategies for improving CRC screening uptake in the practice's patient panel. In cases where the PCP was unavailable, an office staff member was approached. A brief description of the RCT was followed by a semi-structured interview assessing usual practice regarding CRC screening referral and follow up. The direction of the discussion was guided by PCP responses. A variety of resources were provided: a binder with up-to-date scientific evidence about CRC screening recommendations and printed patient education materials, and order forms for refilling supplies. Specific directives were following up to make sure patients had made appointments with a gastroenterologist and offering 3-day FOBT. The detailer attempted to elicit a verbal commitment to do at least one new thing to strengthen the probability that patients would be screened. The TTE was based on the investigators' previously tested model and involved a semi-structured protocol in which the first goals were to build rapport and assess level of knowledge and readiness to be screened. In contrast to the earlier RCT, the current study's TTE clearly represented colonoscopy as the screening method of choice, while encouraging alternative screening methods as well. This emphasis was consistent with goals of the New York City Department of Health and Mental Hygiene and the American Cancer Society at the time of the study. Rapport established, the TTE dialogue focused on identifying and addressing barriers that might impede receipt of screening. Verbal commitments were elicited: to speak with the PCP and make an appointment for a colonoscopy, or request a home stool test, as appropriate. Follow up calls assessed progress towards achieving goals.

Three types of data were collected. Baseline survey data assessed eligibility and measured a variety of demographic and other variables. Implementation data monitored the extent to which the AD and TTE interventions had been conducted as planned. And outcome data (CRC screening one year post-randomization) was based on medical claims data.

ELIGIBILITY:
Inclusion Criteria:

* out of compliance with recommended CRC screening
* having a 'regular doctor' (for women, could be gynecologist)
* stated intention to remain in benefit fund for at least one year
* age 50 to 75
* reachable by telephone
* able to communicate in English
* ability to grant informed consent

Exclusion Criteria:

* colonoscopy in past 10 years
* flexible sigmoidoscopy, barium enema or CT colonography in past 5 years
* stool DNA in past 3 years
* 3 day FOBT or FIT within past year
* history of colorectal polyps, inflammatory bowel disease, irritable bowel syndrome, Crohn's disease, ulcerative colitis, or current treatment for any type of cancer

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2009-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Screening | one year
  defined as colonoscopy, flexibile sigmoidoscopy, barium enema, CT colonography or DNA stool test based on medical claims paid by benefit fund

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Basch, PhD, Principal Investigator — Teachers College, Columbia University

REFERENCES:
- [Derived] Basch CH, Basch CE, Zybert P, Wolf RL. Failure of Colonoscopy Knowledge to Predict Colonoscopy Uptake. J Community Health. 2016 Oct;41(5):1094-9. doi: 10.1007/s10900-016-0194-6. PMID 27098522
- [Derived] Basch CH, Basch CE, Zybert P, Wolf RL. Fear as a Barrier to Asymptomatic Colonoscopy Screening in an Urban Minority Population with Health Insurance. J Community Health. 2016 Aug;41(4):818-24. doi: 10.1007/s10900-016-0159-9. PMID 26831486
- [Derived] Wolf RL, Basch CE, Zybert P, Basch CH, Ullman R, Shmukler C, King F, Neugut AI. Patient Test Preference for Colorectal Cancer Screening and Screening Uptake in an Insured Urban Minority Population. J Community Health. 2016 Jun;41(3):502-8. doi: 10.1007/s10900-015-0123-0. PMID 26585609
- [Derived] Basch CE, Zybert P, Wolf RL, Basch CH, Ullman R, Shmukler C, King F, Neugut AI, Shea S. A Randomized Trial to Compare Alternative Educational Interventions to Increase Colorectal Cancer Screening in a Hard-to-Reach Urban Minority Population with Health Insurance. J Community Health. 2015 Oct;40(5):975-83. doi: 10.1007/s10900-015-0021-5. PMID 25850386